CLINICAL TRIAL: NCT06687239
Title: Does Blind Measurement of Biometric Indices Improve the Accuracy of Fetal Weight Estimation
Brief Title: Blind Measurement in Fetal Weight Estimation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eran Brazilay, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Eran Brazilay, MD PhD, Head of OBGYN ultrasound unit, Assuta Ashdod Hospital
Organization: Assuta Ashdod Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0081-23-AAA
Record Dates: First submitted 2024-10-31; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy
Keywords: estimated fetal weight; Blinded measurements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blinded (Other): Blinded biometric measurements
  Interventions: Diagnostic Test: Blinded estimation of fetal weight
- Non-blinded (Other): Non-blinded biometric measurements
  Interventions: Diagnostic Test: Non blinded estimation of fetal weight

INTERVENTIONS:
Diagnostic Test: Blinded estimation of fetal weight — Blinded ultrasound-based estimation of fetal weight
  Arms: Blinded
Diagnostic Test: Non blinded estimation of fetal weight — Non-blinded ultrasound-based estimation of fetal weight
  Arms: Non-blinded

SUMMARY:
Woman who are expected to give birth in the next 72 hours will be allocated randomly to a study group of blinded measurements for estimated fetal weight and a control group of non-blinded measurements. Accuracy of estimations will be compared between the groups.

DETAILED DESCRIPTION:
Estimating fetal weight using ultrasound is an essential component in fetal medicine and prenatal treatment.

A study that was conducted as a part of the INTERGROWTH-21 project established international standards for fetal growth by documenting 3 measurements of biometry indices, which included head circumference, abdominal circumference, femur length and biparietal diameter (BPD). The measurements were not disclosed to the investigator in order to prevent bias.

In a recent study it was found that use of the average of the 3 biometric measurements compared with a single measurement for the purposes of estimating fetal weight, is more accurate. However, the measurements were disclosed to the investigator.

Currently, no studies have examined whether there blinded measurements are significantly better than non-blinded measurements.

The aim of this study is to compare blinded to non-blinded biometric measurements for estimation of fetal weight.

Woman who are expected to give birth in the next 72 hours will be asked to participate in the study. After singing an informed consent, participants will be randomly allocated to a study group of blinded measurements for estimated fetal weight and a control group of non-blinded measurements. Estimation of fetal weight will be performed using the Hadlock-4 formula in triplicate measurements. In the study group the measurement will be blinded from the sonographer and measurements will be revealed only upon completion of all measurements. In the control group, the same measurements will be conducted without blinding of the measurements during the assessment. Accuracy of estimations will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age between 37 and 41 weeks
* Expected delivery within 72 hours

Exclusion Criteria:

* Major Malformations
* Active labor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Estimated fetal weight accuracy | From estimation of fetal weight to delivery, up to 72 hours.
  Accuracy of fetal weight estimation. A continuous variable, measured as the absolute difference between birthweight and estimated fetal weight in grams.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be shared upon reasonable request

REFERENCES:
- [Background] Sheiman V, Frenkel A, Glick N, Tovbin J, Neeman O, Barzilay E. Ultrasonic Estimation of Fetal Weight: Are Averaged Triplicate Measurements More Accurate Than Single Measurements? J Ultrasound Med. 2024 Nov;43(11):2147-2152. doi: 10.1002/jum.16545. Epub 2024 Aug 6. PMID 39105327
- [Background] Papageorghiou AT, Ohuma EO, Altman DG, Todros T, Cheikh Ismail L, Lambert A, Jaffer YA, Bertino E, Gravett MG, Purwar M, Noble JA, Pang R, Victora CG, Barros FC, Carvalho M, Salomon LJ, Bhutta ZA, Kennedy SH, Villar J; International Fetal and Newborn Growth Consortium for the 21st Century (INTERGROWTH-21st). International standards for fetal growth based on serial ultrasound measurements: the Fetal Growth Longitudinal Study of the INTERGROWTH-21st Project. Lancet. 2014 Sep 6;384(9946):869-79. doi: 10.1016/S0140-6736(14)61490-2. PMID 25209488
- [Background] Chang TC, Robson SC, Spencer JA, Gallivan S. Ultrasonic fetal weight estimation: analysis of inter- and intra-observer variability. J Clin Ultrasound. 1993 Oct;21(8):515-9. doi: 10.1002/jcu.1870210808. PMID 8270670
- [Background] Hammami A, Mazer Zumaeta A, Syngelaki A, Akolekar R, Nicolaides KH. Ultrasonographic estimation of fetal weight: development of new model and assessment of performance of previous models. Ultrasound Obstet Gynecol. 2018 Jul;52(1):35-43. doi: 10.1002/uog.19066. Epub 2018 Jun 3. PMID 29611251
- [Background] Perlow JH, Wigton T, Hart J, Strassner HT, Nageotte MP, Wolk BM. Birth trauma. A five-year review of incidence and associated perinatal factors. J Reprod Med. 1996 Oct;41(10):754-60. PMID 8913978